CLINICAL TRIAL: NCT06644417
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQA3605 Tablets in Treated Subjects With Chronic HBV Infection With Low-level Viremia (LLV)
Brief Title: Clinical Study of TQA3605 Tablets Combined With Nucleoside (Acid) Analogs (NAs) Drugs Compared With NAs Drugs in the Treatment of Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA3605-II-01
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: HBV Infection With LLV
MeSH Terms: interventions — nas

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQA3605 Placebo plus NAs (Placebo Comparator): TQA3605 placebo plus NAs drug was administered for 24 weeks and NAs was continued until 32 weeks
  Interventions: Drug: TQA3605 Placebo plus NAs
- 100mg TQA3605 tablets plus NAs (Experimental): 100mg TQA3605 tablets plus NAs drug was administered for 24 weeks and NAs was continued until 32 weeks
  Interventions: Drug: TQA3605 tablets plus NAs
- 200mg TQA3605 tablets plus NAs (Experimental): 200mg TQA3605 tablets plus NAs drug was administered for 24 weeks and NAs was continued until 32 weeks
  Interventions: Drug: TQA3605 tablets plus NAs

INTERVENTIONS:
Drug: TQA3605 tablets plus NAs — TQA3605 tablets is core protein regulator
  Arms: 100mg TQA3605 tablets plus NAs; 200mg TQA3605 tablets plus NAs
Drug: TQA3605 Placebo plus NAs — Placebo without drug substance
  Arms: TQA3605 Placebo plus NAs

SUMMARY:
This study is a phase II multicenter, randomized, double-blind, placebo controlled study designed to evaluate the efficacy and safety in LLV subjects and demonstrate that TQA3605 tablets combined with oral NAs drugs can improve the efficacy and safety of LLV subjects compared with oral NAs drug.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 (including boundary values), male or female.
* At the time of screening, etiological or clinical or pathological evidence of hepatitis B virus infection has been more than 1 year; HBsAg positive, 10 IU/mL <HBV DNA≤2000 IU/mL, ALT≤3×ULN (upper limit of normal); No obvious cirrhosis was found by the researchers.
* Continuous administration of any nucleoside (acid) analogues for more than 1 year and a stable regimen of ≥6 months prior to screening.
* Able to communicate well with researchers, understand and comply with the requirements of the study, understand and sign the informed consent.
* Male subjects with fertile female partners or female subjects of childbearing age were willing to voluntarily take effective contraceptive measures within 3 months after screening.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or breastfeeding women.
* Co-infection with other viruses such as hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, human immunodeficiency virus, syphilis.
* A history of cirrhosis or evidence of significant fibrosis or cirrhosis at pre-screening/screening time.
* The subject had a history of hepatocellular carcinoma (HCC) before or at the time of screening, or was suspected of HCC.
* A history of malignant tumors within 5 years prior to screening, except for certain cancers that can be completely cured by surgical resection.
* Subjects with other chronic liver diseases, including but not limited to autoimmune liver disease, alcoholic liver disease, and hepatolenticular degeneration.
* Have previously received organ transplantation and bone marrow transplantation.
* Abnormal laboratory examination indicators that do not meet the requirements of the program during screening.
* Poorly controlled thyroid disease, or clinically significant thyroid dysfunction.
* Autoimmune diseases include but are not limited to: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, psoriasis, autoimmune uveitis, etc.;
* In addition to liver disease, there are significant systemic or major diseases, including recent congestive heart failure, unstable coronary heart disease, arterial revasodilation, respiratory disease, digestive disease, renal insufficiency, stroke, transient ischemic attack, organ transplantation, psychiatric disease, etc. Uncontrolled systemic disease: poor blood pressure control; Diabetes has poor blood sugar control.
* Received any systemic antitumor (including radiation) or immunosuppressive therapy (including biological immune inhibitors), or immunomodulatory therapy (including non-biological immunomodulatory oral drugs) in the 6 months prior to screening.
* Receiving high doses of systemic corticosteroids within 3 months prior to the screening period.
* A history of alcohol and drug abuse within 1 year prior to the screening period.
* Blood transfusion ≤2 months before screening and/or blood donation ≤1 month before screening. Note: Participants were not allowed to donate blood throughout the study period.
* Have a history of allergy to the experimental drug or its excipients.
* Participated in clinical trials of hepatitis B core protein allosteric regulators.
* The subject has participated in a clinical trial and received the investigational drug during the period prior to the first administration of the study: 5 half-lives or twice the duration of the biological effect of the study treatment or 90 days (if the half-life or duration is unknown).
* History or status of cardiovascular disease: history of risk factors for tip torsion ventricular tachycardia, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory tests. Family history of long QT syndrome or Brugada syndrome. The Electrocardiogram (ECG) showed clinically significant abnormalities. Heart Rate (HR)≤45 bpm.
* Those that researchers believe should not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
HBV DNA (Hepatitis B virus Deoxyribonucleic Acid) | 24 weeks
  Percentage of subjects with HBV DNA below the lower limit of quantitative detection (<10 IU/mL) at 24 weeks of treatment

SECONDARY OUTCOMES:
Incidence and severity of Adverse events (AEs) | 32 weeks
  The incidence and severity of AEs were determined by changes in physical examination, vital signs, electrocardiogram, and laboratory tests
Incidence and severity of serious adverse events (SAEs) | 32 weeks
  The incidence and severity of SAEs were determined by changes in physical examination, vital signs, electrocardiogram, and laboratory tests
HBV DNA (<10 IU/mL) | Weeks 12, Weeks 16, Weeks 28, Weeks 32
  Percentage of subjects with HBV DNA below the lower limit of quantitative detection (<10 IU/mL)
HBV DNA (<10 IU/mL) | Weeks 12, Weeks 16, Weeks 24, Weeks 28, Weeks 32
  Percentage of subjects with HBV DNA below the lower limit of quantitative detection (<10 IU/mL)
Hepatitis B e antigen (HBeAg) Serology | Weeks 12, Weeks 24, Weeks 32
  Percentage of subjects with HBeAg serologic clearance and/or serologic conversion (for HBeAg positive at baseline only)
Alanine Aminotransferase (ALT) relapse rate | Weeks 12, Weeks 24, Weeks 32
  Renormalize ALT over time in subjects with baseline ALT>upper limit of normal (ULN) in the absence of enzyme-lowering Liver protection medicine
Breakthroughs in virology | Weeks 12, Weeks 24, Weeks 32
  Percentage of subjects with a virological breakthrough
Actual values and changes of HbsAg (Hepatitis B Surface Antigen) | Weeks 12, Weeks 24, Weeks 32
  Actual values and changes of HbsAg over time relative to baseline
Actual values and changes of HBeAg | Weeks 12, Weeks 24, Weeks 32
  Actual values and changes of HBeAg over time relative to baseline
Actual values and changes of HBV DNA | Weeks 12, Weeks 24, Weeks 32
  Actual values and changes of HBV DNA over time relative to baseline
HBV RNA (Hepatitis B virus Ribonucleic Acid) | Weeks 12, Weeks 24, Weeks 32
  Actual values and changes of HBV RNA over time relative to baseline
Actual values and changes of Human Hepatitis B virus core antigen - associated antigen (HbcrAg) | Weeks 12, Weeks 24, Weeks 32
  Actual values and changes of HbcrAg over time relative to baseline
(Cmax, ss) Steady-state maximum concentration | Day 1, Day 29, Day 57, Day 85, Day 113, Day 169
  Steady-state maximum concentration of TQA3605
(Cmin, ss) Steady state minimum concentration | Day 1, Day 29, Day 57, Day 85, Day 113, Day 169
  Steady-state minimum concentration of TQA3605

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical Universitybeijing Institute of Hepatology, Beijing, Beijing Municipality
  - Meng Chao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Zunyi Medical University Affiliated Hospital, Zunyi, Guizhou
  - Zhengzhou No.6 peoples Hospital, Zhengzhou, Henan
  - The Second XIANGYA Hospital Of Central South University, Changsha, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The sixth people's Hospital Of Shenyang, Shenyang, Liaoning
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang